CLINICAL TRIAL: NCT05756231
Title: Cultural and Linguistic Adaptation and Normative Study of the Turkish Version of the Free and Cued Selective Reminding Test: 16-Word Version (FCSRT-T)
Acronym: FCSRT-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Jbid DURSUN UNCU, Clinical Neuropsychologist, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2019/778
Record Dates: First submitted 2023-01-26; First posted 2023-03-06 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Dementia; Memory Impairment
Keywords: Alzheimer Disease; Memory Complaint; Memory; Dementia; Free and Cued Selective Reminding Test; Adaptation; Validity
MeSH Terms: conditions — Dementia; Memory Disorders; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Turkish Adaptation Study of Free and Cued Selective Reminding Test (SIHT-16) (Experimental): Outcomes of Turkish adaptation of Free and cued selective reminding test (SIHT-16) is compared with memory and non-memory test in three alternative lists: a,b, and c parallel lists. The participants are assessed in neurological diagnosis routine.
  Interventions: Behavioral: SIHT-16

INTERVENTIONS:
Behavioral: SIHT-16 — a pencil-paper assessment tool.

SUMMARY:
An Adaptation Study of Free and Cued Selective Reminding Test in Turkish

DETAILED DESCRIPTION:
As very commonly used for objectifying Alzheimer Disease memory deficits, an adaptive selection of word choices are done for the use of free and cued selective reminding test (FCSRT) procedure in Turkish population. In this study the validity and reliability of the test to measure memory deficits in persons with memory complaints will be discussed.

ELIGIBILITY:
Inclusion Criteria:

* having memory complaints
* demanding clinical consultation for the memory complaint

Exclusion Criteria:

* vascular pathology
* extrapyramidal findings
* psychiatric illness
* epilepsy
* cognition affecting drug use

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Validity of translation | once
  Variances of answers given to each form will be compared to each other to know if they are similar or different.
Factor Analyses | once
  Factor Analyses must be conducted to redefine the weight of each item on measuring memory deficits to be sure that turkish words version is similar to original factor weights.
Validity of the ability of the measure to objectify the memory deficit in dementia | once
  Test measures must be sensitive enough to objectify a memory deficits even in early stages of dementia. The scores of memory test in early and late stages of dementia will be compared to see if they are different. It's expected to be different.

CONTACTS AND LOCATIONS:
Overall Officials: İ. Hakan Gürvit, Prof. MD., Study Director — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No